CLINICAL TRIAL: NCT04835311
Title: Retrospective Evaluation of Functional and Sexological Results of Surgical Perineal Repair
Acronym: SEX-RPC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/THESE/RDT-01
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-09

CONDITIONS: Complications; Perineal Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical perineal repair — women who have undergone surgical perineal repair (codes CCAM JMMA002 and/or HKCA005)

SUMMARY:
Vaginal laxity" syndrome is an increasingly frequent reason for gynecological consultations. Patients complain above all of a sensation of excessive vaginal looseness. This syndrome can be isolated or associated with genital prolapse. Women with vaginal laxity may experience sexual dysfunction manifested by hypersensitivity during penetration and vaginal gas, resulting in decreased libido. Among urogynecology patients, vaginal laxity has been reported in up to 24% of cases, with a mean discomfort of 5.7 (on a scale of 0 to 10). Vaginal laxity is more common in younger women who have given birth vaginally. Gynecologic examination usually finds widening of the urogenital hiatus during the Valsalva maneuver, suggesting that vaginal laxity may be a manifestation of hyperdistensibility or disinsertion of the levator ani muscles. Campbell et al. noted that vaginal laxity was reported by 38% of 22621 women attending a urogynecology clinic and was associated with vaginal parity, prolapse symptoms, stress, and urinary urgency incontinence, reduced sensation on the ePAQ-PF questionnaire. In an IUGA survey of member physicians, 83% of respondents felt that vaginal laxity was underreported by patients.

The most common clinical definition of vaginal laxity is a urinary meatus to vulvar fork distance (GH measure of the POP-Q classification) > or = 4cm.

The first-line treatment for vaginal laxity is perineal rehabilitation. If this fails, surgical perineal repair, combining posterior perineorrhaphy and myorrhaphy of the pubo-rectal bundles of the levator ani muscles, can be performed with the aim of narrowing the introital vaginal caliber and improving the symptoms of laxity. This procedure is poorly evaluated in the literature.

The purpose of this study is to evaluate the functional and sexological results of surgical perineal repair.

ELIGIBILITY:
Inclusion Criteria:

* women who underwent surgical perineal repair (CCAM codes JMMA002 and/or HKCA005) between July 2012 and September 2020 at Nîmes University Hospital.
* Adult patient (≥18 years old)
* Enrolled in a social security plan
* Patient does not object to the study

Exclusion Criteria:

* Prolapse surgery without perineal repair
* Perineal repair without levator myorrhaphy
* Patient who objected to the use of their data.
* Pregnancy since the operation
* Persons under court protection,
* Person participating in another research study with an ongoing exclusion period,
* Severely impaired physical and/or psychological health that, in the opinion of the investigator, may affect the participant's compliance with the study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All women who underwent surgical perineal repair (CCAM codes JMMA002 and/or HKCA005) between July 2012 and September 2020 at Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the sexological results of surgical perineal repair. | Day 30
  Validated questionnaire (Pelvi-Perineal Surgery Sexuality Questionnaire). Sexual health = score minimum 2 / maximum 29 (29 = very good sexual health) Discomfort and pain = score minimum 0 / maximum 15 (15 = important discomfort or pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al Salehi A, Zemmache MZ, Allegre L, Fatton B, de Tayrac R. Functional and sexual outcomes following surgical vaginal introital reduction. Prog Urol. 2023 Jul;33(7):370-376. doi: 10.1016/j.purol.2023.05.003. Epub 2023 May 30. PMID 37263901